CLINICAL TRIAL: NCT06704737
Title: Dichoptic Augmented Reality (AR) Training Versus Patching in Adults With Unilateral Amblyopia
Brief Title: AR Training in Adults With Unilateral Amblyopia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EENTAR20230225
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Amblyopia Unilateral; Amblyopia Functional
Keywords: Adult; Augmented reality training; Patching; Neural deficit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR training group (Experimental): Dichoptic augmented reality training with dual-pathway (parvocellular pathway and magnocellular pathway) and interocular push-pull paradigms developed based on neural deficits in adults with unilateral amblyopia.
  Interventions: Device: AR training
- Patching group (Active Comparator): Conventional patching therapy.
  Interventions: Device: Patching

INTERVENTIONS:
Device: AR training — Dichoptic augmented reality training with dual-pathway (parvocellular pathway and magnocellular pathway) and interocular push-pull paradigms developed based on neural deficits in adults with unilateral amblyopia
  Arms: AR training group
Device: Patching — Conventional patching therapy.
  Arms: Patching group

SUMMARY:
This is a single-center, non-randomized controlled trial to compare the effectiveness of binocular AR training with patching for the treatment of adults with unilateral amblyopia.

Specific Aim 1 (Primary): To compare the improvement of visual acuity in the amblyopic eye between AR training and patching for the treatment of adults with unilateral amblyopia.

Specific Aim 2 (Secondary): To compare the changes of visual functions and pathway selective neural activity in the early visual and cortex subcortical nuclei including the lateral geniculate nucleus between AR training and patching for the treatment of adults with unilateral amblyopia.

DETAILED DESCRIPTION:
Patching the fellow eye (FE) is typically the first line of amblyopia therapy. Patching treatment has been thought to be effective only when started before the age of eight and might bring limited benifits for adults who have decreased visual cortex plasticity (Bhola et al., 2006). However, recent animal and human studies have demonstrated that visual cortex plasticity and visual functions can be enhanced later in life (Kind et al., 2002; Pineles et al., 2020), paving the way for new strategies for amblyopia treatment.

Dichoptic/binocular digital therapy has been developed with hope to improve visual functions in amblyopia post the critical period. However, no widely accepted binocular treatments with superiority to patching is available in adults with unilateral amblyopia (Pineles et al., 2020; Oscar et al., 2023). Here, we designed an innovative binocular therapy using augmented reality (AR) training, based on neural deficits in amblyopia, in order to achieve better outcomes.

Selective deficits were found in the parvocellular pathway (P pathway) compared to the magnocellular pathway (M pathway) in the monocular processing of visual information in the amblyopic eye (AE) (Wen et al., 2021). In addition to monocular deficits, imbalanced binocular suppression may also play important roles in the visual deficits of amblyopia as suggested by clinical evidence (DeSantis, 2014; Von Noorden, 1996) and psychophysical studies (Baker et al., 2008; Holopigian et al., 1988; Li et al., 2011; Zhou et al., 2013). Based on the neural deficits in unilateral amblyopia, we first apply the push-pull approach (Xu, He & Ooi, 2010; Ooi et al., 2013), which was aimed to reduce sensory eye dominance in previous literatures, into the rebalance of functions of M and P pathways in the AE and the rebalance of binocular interaction, to improve the high spatial detail perception of the AE in daily life under binocular viewing condition, as well as binocular functions.

Using AR technique combined with dichoptic device, images are processed differently and dichopticaly presented to each eye of the patients in real time, same in the content but different in contrast, spatial frequency, temporal frequency, and signal-to-noise ratio, allowing them to interact with the surrounding environment in real time during the visual training. We aim to achieve push-pull in monocular M-P pathways in the AE and interocular P-P pathways in the FE and the AE, in order to selectively improve the function of the P pathway in the AE under binocular viewing condition.

The proposed trial will be conducted in one study sites in China. For the AR training group, patients need to perform AR training for 2 hours per day at home. For the patching group, patients need to patch the FE for 2 hours per day at home.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 years (including 18 years and 50 years);
2. Best-corrected visual acuity worse than 20/30 but no worse than 20/200 in the amblyopic eye, interocular difference of 2 or more lines, with the better eye within the normal range;
3. Patients with deprivation amblyopia should have relieved the deprivation factors such as opacification of the ocular media (e.g. cataract, nonclearing vitreous opacity, corneal opacities) or other occlusion of the visual axis (e.g. blepharoptosis).
4. Normal binocular alignment including strabismic amblyopia with orthotropia after optical refractive correction or surgical correction, or intermittent exotropia within a range of -15 to 0 prism diopters measured by the prism cover test.
5. Patients should have been applyng optical refractive correction for more than 3 months before enrollment.

Exclusion Criteria:

1. Organic eye diseases preventing the establishment of good vision (e.g. ptosis, media opacity, nystagmus, paracentral fixation, acute inflammation like keratitis, optic nerve diseases like glaucoma, retinal diseases);
2. Lesions of the brain preventing the establishment of good vision (e.g. cortical visual impairment);
3. A history of ocular surgery (except strabismus surgery) affecting vision (e.g. retinal detachment repair);
4. A history of ocular trauma affecting vision;
5. Receiving amblyopia therapy (except wearing refractive correction glasses) within 2 weeks before enrollment;
6. History of epilepsy or mental illness, or cognitive defects;
7. Currently taking medications or needing to take medications during the study period that may affect vision;
8. Contraindications to magnetic resonance imaging such as implantable electronic device, metal implants (e.g. metal dentures, craniofacial titanium plates), claustrophobia and pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity at far | 1 week, 1month, 3month, 6month
  Best-corrected visual acuity in the amblyopic eye measured at the distance of 2.5 meters using standardized logMAR visual charts.

SECONDARY OUTCOMES:
Change in visual acuity at near | 1 week, 1month, 3month, 6month
  Best-corrected visual acuity in the amblyopic eye measured at the distance of 2.2 meters using the Freiburg Visual Acuity test.
Change in visual acuity with single tumbling E | 1 week, 1month, 3month, 6month
  Best-corrected uncrowded and crowded visual acuity in the amblyopic eye measured at the distance of 30 centimeters.
Change in contrast sensitivity | 1 week, 1month, 3month, 6month
  Contrast sensitivity in each eye measured with forced-choice test under binocular viewing.
Change in faxation stability | 1 week, 1month, 3month, 6month
  Fixation stability in each eye measured with EyeLink 1000.
Change in binocular phase combination | 1 week, 1month, 3month, 6month
  Binocular integration measured with phase combination test .
Change in binocular rivalry ratio | 1 week, 1month, 3month, 6month
  Binocular rivalry ratio measured with binocular rivalty test
Change in stereopsis | 1 week, 1month, 3month, 6month
  Near stereopsis measured with Titmus Fly Stereotest pattern.
Change in neural activity corresponding to visual inputs in SSVEP | 1 week, 1month, 3month, 6month
  Pathway-selective neural activity in the early visual cortex revealed by SSVEP.
Change in neural activity corresponding to visual inputs in fMRI | 1 week, 1month, 3month, 6month
  Pathway-selective neural activity in the early visual cortex and subcortical nuclei including lateral geniculate nucleus revealed by fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wen, MD, PhD, Study Chair — Eye & ENT Hospital of Fudan University, Shanghai, China
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.

REFERENCES:
- [Result] Ooi TL, Su YR, Natale DM, He ZJ. A push-pull treatment for strengthening the 'lazy eye' in amblyopia. Curr Biol. 2013 Apr 22;23(8):R309-10. doi: 10.1016/j.cub.2013.03.004. PMID 23618663
- [Result] Xu JP, He ZJ, Ooi TL. Effectively reducing sensory eye dominance with a push-pull perceptual learning protocol. Curr Biol. 2010 Oct 26;20(20):1864-8. doi: 10.1016/j.cub.2010.09.043. Epub 2010 Oct 14. PMID 20951044
- [Result] Zhou J, Huang PC, Hess RF. Interocular suppression in amblyopia for global orientation processing. J Vis. 2013 Apr 22;13(5):19. doi: 10.1167/13.5.19. PMID 23608341
- [Result] Li J, Thompson B, Lam CS, Deng D, Chan LY, Maehara G, Woo GC, Yu M, Hess RF. The role of suppression in amblyopia. Invest Ophthalmol Vis Sci. 2011 Jun 13;52(7):4169-76. doi: 10.1167/iovs.11-7233. PMID 21447685
- [Result] Holopigian K, Blake R, Greenwald MJ. Clinical suppression and amblyopia. Invest Ophthalmol Vis Sci. 1988 Mar;29(3):444-51. PMID 3343099
- [Result] Baker DH, Meese TS, Hess RF. Contrast masking in strabismic amblyopia: attenuation, noise, interocular suppression and binocular summation. Vision Res. 2008 Jul;48(15):1625-40. doi: 10.1016/j.visres.2008.04.017. Epub 2008 Jun 10. PMID 18547600
- [Result] Von Noorden GK. Binocular vision and ocular motility. Theory and Management of Strabismus. 1996.
- [Result] DeSantis D. Amblyopia. Pediatr Clin North Am. 2014 Jun;61(3):505-18. doi: 10.1016/j.pcl.2014.03.006. Epub 2014 Apr 14. PMID 24852148
- [Result] Wen W, Wang Y, Zhou J, He S, Sun X, Liu H, Zhao C, Zhang P. Loss and enhancement of layer-selective signals in geniculostriate and corticotectal pathways of adult human amblyopia. Cell Rep. 2021 Dec 14;37(11):110117. doi: 10.1016/j.celrep.2021.110117. PMID 34910903
- [Result] Cruz OA, Repka MX, Hercinovic A, Cotter SA, Lambert SR, Hutchinson AK, Sprunger DT, Morse CL, Wallace DK; American Academy of Ophthalmology Preferred Practice Pattern Pediatric Ophthalmology/Strabismus Panel. Amblyopia Preferred Practice Pattern. Ophthalmology. 2023 Mar;130(3):P136-P178. doi: 10.1016/j.ophtha.2022.11.003. Epub 2022 Dec 14. No abstract available. PMID 36526450
- [Result] Pineles SL, Aakalu VK, Hutchinson AK, Galvin JA, Heidary G, Binenbaum G, VanderVeen DK, Lambert SR. Binocular Treatment of Amblyopia: A Report by the American Academy of Ophthalmology. Ophthalmology. 2020 Feb;127(2):261-272. doi: 10.1016/j.ophtha.2019.08.024. Epub 2019 Oct 13. PMID 31619356
- [Result] Kind PC, Mitchell DE, Ahmed B, Blakemore C, Bonhoeffer T, Sengpiel F. Correlated binocular activity guides recovery from monocular deprivation. Nature. 2002 Mar 28;416(6879):430-3. doi: 10.1038/416430a. PMID 11919632
- [Result] Bhola R, Keech RV, Kutschke P, Pfeifer W, Scott WE. Recurrence of amblyopia after occlusion therapy. Ophthalmology. 2006 Nov;113(11):2097-100. doi: 10.1016/j.ophtha.2006.04.034. PMID 17074568